CLINICAL TRIAL: NCT03699280
Title: Virtual Reality as a Distraction Technique for Management of Acute Pain at Outpatient Hysteroscopy.
Brief Title: Virtual Reality and Outpatient Hysteroscopy
Acronym: VISTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18IC4481
Record Dates: First submitted 2018-09-19; First posted 2018-10-09 (Actual); Results first posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2022-05

CONDITIONS: Acute Pain; Hysteroscopy
Keywords: virtual reality, hysteroscopy, acute pain, distraction technique
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: The study is a randomised control trial involving mixed methods of qualitative and quantitative analysis. The study will include 40 patients attending the outpatient hysteroscopy clinic and randomised to either a VR intervention group or standard procedure by computer-generated randomisation.
  All patients will fill in a questionnaire before and after the procedure. Patients who have been randomised to the VR arm will have a semi-structured interview regarding their experience with VR.
  The clinician performing the procedure will fill in a questionnaire per patient regarding the ease of the procedure and perceived pain levels of the patient. The Clinician performing the procedure and nursing staff's perception regarding feasibility of using the VR equipment for each patient who had the intervention was also assessed through the questionnaire.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): VR video to be played during the procedure
  Interventions: Other: Virtual Reality
- Standard Procedure (No Intervention): Routine protocol outpatient hysteroscopy

INTERVENTIONS:
Other: Virtual Reality — Oculus Go VR device
  Arms: Virtual Reality

SUMMARY:
TITLE Virtual Reality (VR) as a Distraction technique for management of acute pain at Outpatient Hysteroscopy DESIGN Randomised Control Trial (RCT) with Mixed methods - Qualitative and quantitative AIMS To study the role of distraction techniques for management of acute pain in Outpatient Hysteroscopy and to assess feasibility of using Virtual Reality for managing pain.

Primary objective:

• Feasibility of using virtual reality as a distraction technique in management of acute pain in patients undergoing Outpatient Hysteroscopy.

Secondary objectives:

* Understanding the acceptability and effectiveness of VR interventions within the procedural groups and how these might vary as a function of different patient demographics.
* Understanding the factors that might influence the willingness of patients to participate in a future formal trial of the technology.
* Understanding how best to implement the technology and designing of the contents of the VR intervention.
* Understanding the effective mechanisms for the analgesic effect of VR and explore how this could be tailored to individual patients.

POPULATION Patients attending the Outpatient Hysteroscopy clinics ELIGIBILITY Patients undergoing Outpatient Hysteroscopy DURATION 6 months

DETAILED DESCRIPTION:
INTRODUCTION

BACKGROUND Performing procedures for investigation and treatment of gynaecological conditions in the office setting is becoming commonplace. Outpatient gynaecological procedures can reduce risks of general anaesthetic, decrease health care costs and make the procedure more convenient for the patient and provider. However, ensuring adequate pain relief and allaying anxiety during the procedure can prove to be challenging. Appropriate patient selection, counselling and adequate pain management during the procedure can improve patient experience and reduce the number of failed procedures.

Common office gynaecological procedures include outpatient hysteroscopy, colposcopy and large loop excision of transformation zone, manual vacuum aspiration for treatment of miscarriages, intrauterine contraceptive device insertion, hysteroscopic sterilisation and endometrial biopsy.

Pain in gynaecological procedures can originate from the cervix and uterus. The uterine fundus is innervated by sympathetic fibres from T10 to L2, which enter through the uterosacral ligaments via the inferior hypogastric plexus, and by nerves from the ovarian plexuses at the cornua. Parasympathetic fibres from S2 to S4 travel through the broad ligament to enter the cervix at the 3 0 clock and 9 o clock positions to provide innervation to the upper vagina, cervix and the lower uterine segment. The pudendal nerve (S 2,3, 4) supplies the lower vagina and vulva.

Physical, psychological and social factors influence the intensity of pain experienced. Counselling the patients pre procedurally helps to better manage expectations and pain.

Outpatient hysteroscopy is usually performed for patients having abnormal uterine bleeding and subfertility. Pain levels during this procedure can be influenced by the diameter of the hysteroscope. Mini hysteroscopes with an outer diameter of 3.5 mm have been associated with lower pain scores. Additional procedures performed (like polypectomy or Coil insertions) could increase the duration of the procedure and the pain experienced during the procedure. Pain scores in the vaginoscopic approach have been noted to be 3.8 when compared to 5.3 in the traditional group, which uses a speculum and tenaculum.

Pain in hysteroscopy is significantly related to the presence of cervical synechiae, to the duration of the procedure, and to the use of normal saline; conversely, parity seems to have a protective role.

Previous vaginal deliveries, experience of the operator and quicker operative time are known to be associated with successful outcomes of the outpatient procedures. However, nulliparity, postmenopausal status, anxiety and anticipated pain and a history of dsymenorrhoea are known to be associated with higher perception of pain and reduced success rates.

The type of pain relief offered can include various levels of sedation, local anaesthetic, analgesics and verbal support techniques through distraction by conversation, gentle language, music, guided imagery and positive suggestion. A Cochrane Review showed no consistent good quality evidence of a significant difference in safety or effectiveness between different types of pain relief compared with each other or with placebo/ no treatment. There is no consensus on the choice of analgesia for outpatient hysteroscopy and rescue analgesia in the form of intracervical blocks is often used.

In the United Kingdom, most units offer analgesics either as Non Steroidal Anti Inflammatory Drugs (NSAIDs), acetaminophen or oral opiods. NSAIDS such as ibuprofen decrease uterine activity and pain by inhibiting cyclooxygenase and thereby reduce circulating prostaglandins. They reduce pain levels especially postoperatively. Acetaminophen also inhibits the enzyme cyclooxygenase, but its action is in the central nervous system rather in the periphery. Hence is inferior to NSAIDS but is offered to women who cannot tolerate NSAIDS. Oral opiods act by interacting with endogenous opioid mu receptors.

The only pharmacological method that has demonstrated its effectiveness in reducing pain during and 30 minutes after hysteroscopy in several meta-analysis and reviews is paracervical block. However, it fails to anaesthetise the uterus for intrauterine procedures and a previous Cochrane review was unable to confirm this. The administration of the local anaesthetic itself may be uncomfortable, have side effects due to toxicity, may cancel the beneficial effect of performing a vaginoscopic hysteroscopy and does not anaesthetise the uterus. Addition of soda bicarbonate as a buffering agent to the local anaesthetic and using dental syringes with a 27-gauge needle has been seen to decrease the pain during the injection. Topical local anaesthetics on the cervix in the form of gel or sprays have not been shown to be effective.

Women undergoing outpatient hysteroscopy experience significant levels of preoperative anxiety which is higher than patients attending the gynaecology clinic and comparable to those experienced before major surgery under general anaesthesia.

Anxiolytics help reduce anxiety, however they do not have a direct analgesic effect.

Units often employ a trained person to engage with the patient to provide emotional support during the procedure.

Distraction Techniques Type of distraction techniques range from active distraction techniques to passive techniques. Active distraction included interactive toys, virtual reality, guided imagery and relaxation and controlled breathing. Passive distraction techniques included auditory distraction in the form of music and audio-visual distraction through watching television. Intraoperative pain and anxiety rating have been noted to be lower by use of simple intraoperative distraction techniques e.g. interacting with nurses, watching Digital Video Discs or using stress balls.

There has been limited research done on the role of distraction techniques in pain management in outpatient gynaecological procedures. Music has been used as a complementary method to control anxiety and reduce perception of pain by relaxing the patient and causing less discomfort during outpatient hysteroscopy. . However, a RCT showed no positive effect of music on patients' level of pain, anxiety or satisfaction of patient or doctor for office hysteroscopy and colposcopy. Watching the procedure on the screen at office hysteroscopy has not been shown to reduce pain scores.

Women with high level of preprocedural state- trait anxiety are more likely to perceive higher levels of pain and discomfort during colposcopy. Simple passive visual distraction during colposcopic examination was associated with a reduction in pain scores, however anxiety levels were unchanged. A Cochrane review in 2007 concluded that anxiety appears to be reduced by playing music during colposcopy. Although information leaflets did not reduce anxiety levels, they did increase knowledge levels and helped with consenting for the procedure.

Virtual reality is a relatively new intervention, which has been studied as a non-pharmacological method for pain relief. VR as a form of managing pain has been studied in paediatrics, dentistry, burns treatment, treatment of chronic pain. It has not been studied in the management of pain of gynaecological procedures, which are increasingly being performed as office procedures.

It acts as a method of distraction for pain relief by changing the activity of the body's pain modulation system. This multisensory technology gives an immersive and engaging experience and serves as a distraction technique. Head tracking systems, visually stimulating scenery and audio and tactile feedback enable integration of many sensory experiences. Different psychological factors influence the effectiveness of the analgesic effect of VR. While sense of presence influence the effectiveness of VR as a distraction tool, anxiety as well as positive emotions directly affects the experience of pain.

VR distraction has been associated with significant increases in pain threshold and pain tolerance and significant decreases in pain intensity, time spent thinking about pain, and self-reported anxiety, relative to baseline. Repeated exposure did not appear to affect the benefits of VR. Simultaneous exposure to VR and supplementary sound increases pain tolerance.

Pain management in ambulatory procedures should be multimodal and should include both pharmacological and non-pharmacological interventions. Giving the patient a range of options will increase the number of successful procedures in the outpatient setting and improve patient experience.

RATIONALE FOR CURRENT STUDY

To study the role of distraction techniques for management of acute pain in ambulatory gynaecology procedures and to assess feasibility of using Virtual Reality for managing pain.

ASSESSMENT AND FOLLOW-UP

The study will aim to recruit 40 patients and randomise them via computer generated random number allocation to either the VR intervention group or those having treatment as per routine protocol.

Both groups of patients will fill a pre and post procedural questionnaire. Pain and anxiety scores prior to the procedure and after the procedure will be compared against a control group of 20 patients for pain management by standard protocol. Scores will be measured by a Numeric Rating Scale (NRS) which is a validated measure of pain which is easy to use, has high compliance rates and is detects meaningful changes in pain. The NRS is an 11-point scale consisting of integers from 0 through 10; 0 representing ''No pain'' and 10 representing ''worst imaginable pain.'' Respondents select the single number that best represents their pain intensity. Ratings of pre-operative anxiety were measured by an 11-point numeric rating scale: 'How would you rate any anxiety you may currently be feeling' 0 (no anxiety) and 10 (worst anxiety imaginable).

The VR intervention will involve watching a standard content of the video on a mobile device using a VR headset to distract them during the procedure. The duration of the video will be 15 minutes; but the video will only be played for the duration of the outpatient hysteroscopy. Patients are allowed to stop viewing the video if they so desire and this will be recorded.

A semi-structured interview will be conducted with the patients who have received the VR intervention, each lasting approximately 20 minutes. The semi structured interviews will allow for all participants to be asked similar question within a flexible framework. The interviews will be conducted within 30 minutes of the procedure, in a suitable location and will be recorded on a digital voice recorder. The questions will be focused on the women's experiences of the procedure, in specific pain perception and questions around the VR intervention as well as any other aspect of their hospital care they felt to be relevant. If further clarification or exploration of any particular aspect of their care was required, the interview will readdress these topics before the end of the interview. Interviews will continue until no new information was being obtained, indicating that the theoretical saturation point had been reached.

Clinician and nursing staff's perception regarding feasibility of using the VR equipment was also assessed through a questionnaire. The clinician questionnaire will also assess the ease of the procedure and perceived pain scores for the patient.

Patient follow up will not be routinely arranged for the purpose of the study. Routine follow up as per clinical requirements will be arranged as routine for the procedure performed.

The study will end once the proposed numbers of patients have been recruited and data analysis completed. Participants will be debriefed after their participation in the study and will be directed to suitable support agencies if necessary.

STATISTICS AND DATA ANALYSIS

The recruitment of women and interviewing proceeded alongside data coding and preliminary analysis.

Interviews will be transcribed verbatim and initially coded by reading and re reading the transcript and making notes, drawing on the observations made during the interviews and transcription. Transcripts will be coded line-by-line, describing, summarising and attending to linguistic elements such as pronoun and metaphor use. The transcripts will be entered into a qualitative software package (N6) and a thematic analysis undertaken from the emergent themes developed from these codes and cluster with related themes. Initial coding is Initial phase will involve open coding. Axial coding and selective coding with use of constant comparison will enable a cyclical and iterative process on the principles of grounded theory. Analytic frame for the analysis will be linked to the primary and secondary aims.

The statistically analysis with include statistical comparison of pre and post anxiety and pain scores as a function of membership of VR or control groups. Analysis of covariance (ANCOVA) will be used to determine whether the VR intervention led to a significantly difference between baseline and follow up pain and anxiety scores between VR and control arm.

Staff questionnaires will be analysed to correlate pain scores of actual vs. perceived and feasibility of carrying out the intervention will be assessed.

Demographic data would include age, parity, menopausal status and ethnicity. Data and all appropriate documentation will be stored for a minimum of 10 years after the completion of the study, including the follow-up period.

REGULATORY ISSUES

ETHICS APPROVAL The Chief Investigator has obtained approval from the Newcastle and North Tyneside 1 National Research Ethics Committee..The study must be submitted for Site Specific Assessment (SSA) at each participating National Health Service (NHS) Trust. The Chief Investigator will require a copy of the Trust Research &Development approval letter before accepting participants into the study. The study will be conducted in accordance with the recommendations for physicians involved in research on human subjects adopted by the 18th World Medical Assembly, Helsinki 1964 and later revisions.

CONSENT Consent to enter the study will be sought from each participant only after a full explanation has been given, an information leaflet offered and time allowed for consideration. Signed participant consent will be obtained. The right of the participant to refuse to participate without giving reasons will be respected. After the participant has entered the study the clinician remains free to give alternative treatment to that specified in the protocol at any stage if he/she feels it is in the participant's best interest, but the reasons for doing so will be recorded. In these cases the participants remain within the study for the purposes of follow-up and data analysis. All participants are free to withdraw at any time from the protocol treatment without giving reasons and without prejudicing further treatment.

In the event of the patient and the staff nurse consenting for the study but the gynaecologist not consenting for the procedure, the patient will be recruited and randomised as per protocol. In the event of the patient and the gynaecologist consenting for the study, but the staff nurse not consenting for the procedure, the patient will be recruited and randomised as per protocol. In these instances, the staff nurse and / or the gynaecologist will not fill the questionnaire and a note will be made.

CONFIDENTIALITY

Confidentiality Information related to participants will be kept confidential and managed in accordance with the Data Protection Act, NHS Caldecott Principles, The Research Governance Framework for Health and Social Care, and the conditions of Research Ethics Committee Approval.

- Record Retention and Archiving When the research trial is complete, the records are kept for a further 10 years. The approved repository for long-term storage of local records is the Trust Modern Records Centre

The Chief Investigator will preserve the confidentiality of participants taking part in the study and is registered under the Data Protection Act.

INDEMNITY Imperial College London holds negligent harm and non-negligent harm insurance policies that apply to this study.

SPONSOR Imperial College London will act as the main Sponsor for this study. Delegated responsibilities will be assigned to the NHS trusts taking part in this study.

FUNDING The study is a part of an MSc (Master of Science) thesis and there is no funding this study.

8.7 AUDITS The study may be subject to inspection and audit by Imperial College London under their remit as sponsor and other regulatory bodies to ensure adherence to GCP (Good Clinical Practice) and the NHS Research Governance Framework for Health and Social Care (2nd edition).

STUDY MANAGEMENT

The day-to-day management of the study will be co-ordinated through Nandita Deo, Consultant Obstetrician and Gynaecologist and PI for the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients: Inclusion criteria will include all women of at least 18 - 70 years of age, planned for an office hysteroscopy.

Staff: Inclusion criteria will include the clinician performing the outpatient hysteroscopy and the nurse supporting the clinic.

Exclusion Criteria:

Patients:

* Hearing impairments and blindness
* Any known anatomical characteristics that may make performing the office procedure more difficult (e.g., cervical conization, Manchester Fothergill).
* The denial or withdrawal of oral informed consent Staff: The denial or withdrawal of informed consent

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2018-08-04 (Actual); Primary Completion 2018-10-06 (Actual); Study Completion 2018-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nandita Deo, FRCOG, Principal Investigator — Imperial College London
Locations (1):
- Whipps Cross University Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan E, Foster S, Sambell R, Leong P. Clinical efficacy of virtual reality for acute procedural pain management: A systematic review and meta-analysis. PLoS One. 2018 Jul 27;13(7):e0200987. doi: 10.1371/journal.pone.0200987. eCollection 2018. PMID 30052655
- [Result] Deo N, Khan KS, Mak J, Allotey J, Gonzalez Carreras FJ, Fusari G, Benn J. Virtual reality for acute pain in outpatient hysteroscopy: a randomised controlled trial. BJOG. 2021 Jan;128(1):87-95. doi: 10.1111/1471-0528.16377. Epub 2020 Jul 22. PMID 32575151

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitments as defined in the protocol
Period: Overall Study
Arm/Group | Virtual Reality | Standard Procedure
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Reality | Standard Procedure | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (5.2) | 31.1 (5.4) | 31.2 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 20 | 20 | 40
Menopausal Status [Count of Participants; unit: Participants]
  Pre-menopausal | 7 | 7 | 14
  Post-menopausal | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Worst Pain Scores
Description: This outcome measure assessed the feasibility of using virtual reality as a distraction technique in the management of acute pain in patients undergoing Outpatient Hysteroscopy.
  'Worst pain scores' indicated the most pain experienced during the procedure, even if momentary. It was based on a numeric rating score (11-point scale from 0 to 10; 0 representing 'no pain' and 10 representing 'worst imaginable pain'). The outcome value refers to the worst pain experienced by the participant during the Hysteroscopy procedure.
Time Frame: during the hysteroscopy procedure, an average of 10 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality | Standard Procedure
Number analyzed (Participants) | 20 | 20
score on a scale | 5.65 (2.4) | 7.85 (2.56)

2. Primary Outcome: Average Pain Scores
Description: This outcome measure assessed the average pain experienced by the participants during the hysteroscopy procedure with virtual reality intervention. The pain scores were based on numeric rating scores (11-point scale from 0 to 10; 0 representing 'no pain' and 10 representing 'worst imaginable pain').
  Data from the two time points in the time frame were combined and calculated as an average.
Time Frame: 10 minutes immediately before and after the procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality | Standard Procedure
Number analyzed (Participants) | 20 | 20
score on a scale | 3.7 (2.66) | 6 (2.62)

3. Primary Outcome: Anxiety Scores
Description: Anxiety scores were measured on a numeric rating score (scale of 0-10, with 0 representing 'no anxiety' and 10 representing 'worst imaginable anxiety'). The anxiety scores measured during the procedure were reported in this outcome measure.
Time Frame: during the hysteroscopy procedure, an average of 10 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality | Standard Procedure
Number analyzed (Participants) | 20 | 20
score on a scale | 3.33 (2.03) | 5.45 (3.35)

ADVERSE EVENTS:
Time Frame: Data collection for adverse events was during when the intervention was administered - i.e. during the procedure and immediately afterwards, an average of 10 minutes.
Arm/Group | Virtual Reality | Standard Procedure
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT03699280/Prot_SAP_000.pdf